CLINICAL TRIAL: NCT02086292
Title: The Influence of Lidocaine Volume on Discomfort During Administration of Local Anesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/2297D
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Needlestick Injuries
Keywords: Injections; Lidocaine; Pain; Healthy volunteers
MeSH Terms: conditions — Needlestick Injuries; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 milliliter lidocaine (Experimental): 2 ml 1% Lidocaine in one ring finger, 1 ml 2% Lidocaine in the other ring finger
  Interventions: Procedure: 2 ml 1% Lidocaine
- 1 milliliter lidocaine (Experimental): 1 ml 1% Lidocaine in one ring finger, 2 ml 2% Lidocaine in the other ring finger
  Interventions: Procedure: 1 ml 2% Lidocaine

INTERVENTIONS:
Procedure: 2 ml 1% Lidocaine
  Arms: 2 milliliter lidocaine
Procedure: 1 ml 2% Lidocaine
  Arms: 1 milliliter lidocaine

SUMMARY:
The aim of the study is to find a simple method for pain reduction that can be used in clinical practice when administering digital nerve block with a single subcutaneous injection. It will be investigated whether a smaller volume of lidocaine can decrease pain during injection.

DETAILED DESCRIPTION:
Healthy volunteers will receive a single subcutaneous injection digital nerve block at the base of each ring finger. 2ml 1% lidocaine in one of the fingers, and 1 ml 2% lidocaine in the other. After each injection, the subject will be asked to evaluate the pain on a visual analog scale (0-100 mm). Additionally the sensibility will be tested with a Semmes-Weinstein monofilament, to evaluate if the different methods achieve desired anesthetic effect.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 65

Exclusion Criteria:

* regular use of analgesics
* known hypersensitivity of local anaesthetic
* renal-, heart- or liver disease
* known peripheral neuropathy or diabetes mellitus
* local infection on injection site
* circulation disorders in upper extremities (e.g. Raynaud´s phenomenon)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pain | 60 seconds
  1. visual analog scale 0-100mm
  2. questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, prof md, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of neuroscience, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Ballo S, Hjelseng T, Tangen LF, Lundbom JS, Skarsvag T, Finsen V. The Influence of Injected Volume on Discomfort During Administration of Digital Block. J Hand Surg Asian Pac Vol. 2016 Oct;21(3):369-73. doi: 10.1142/S2424835516500363. PMID 27595956